CLINICAL TRIAL: NCT07297004
Title: Stereotactic Body Radiation Therapy for Unresectable Locally Recurrent Rectal Cancer: A Prospective, Single-arm, Phase II Study
Brief Title: Stereotactic Body Radiation Therapy for Unresectable Locally Recurrent Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT-ULRRC
Record Dates: First submitted 2025-02-13; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Unresectable Locally Recurrent Rectal Cancer
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): SBRT for unresectable locally recurrent rectal cancer
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — SBRT for unresectable locally recurrent rectal cancer

SUMMARY:
Research Objectives and Principles: Through a prospective study, explore the effectiveness and safety of stereotactic body radiation therapy (SBRT) in the treatment of unresectable locally recurrent rectal cancer (ULRRC), providing high-level evidence for the use of SBRT in ULRRC treatment.

Primary Objective: R0 resection rate. Secondary Objectives: 1-year local progression-free survival (LPFS) and overall survival (OS), 2-year LPFS and OS, and side effects of the treatment.

Study Design: A single-arm, open-label, prospective phase II study. Study Population and Expected Enrollment: Patients with unresectable locally recurrent rectal adenocarcinoma, with an expected enrollment of 20 patients.

Scheduled Visits and Duration: December 2024 to November 2026. Trial Duration: December 2024 to November 2026. Intervention: SBRT for unresectable locally recurrent rectal cancer. Statistical Hypothesis: Enrolled patients are those with unresectable recurrent rectal cancer. Based on previous literature reports and retrospective clinical data from our center, it is hypothesized that the R0 resection rate for patients with unresectable locally recurrent colorectal cancer who do not receive SBRT is 20%, while the R0 resection rate for those receiving SBRT intervention is 50%. Using Simon's optimal two-stage study design, a single-arm study, with α set at 0.05 and 1-β at 0.80, and an expected loss to follow-up rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. 18-75 years of age;
3. Histologically, cytologically, or radiologically confirmed tumor recurrence, and the MDT assesses that the recurrent lesion cannot achieve R0 resection (unresectable defined as: 1) Pelvic MRI shows infiltration of S2 or above, 2) and/or lateral pelvic invasion, 3) and/or neurovascular invasion of the pelvic, 4) No indication for R0 resection after MDT discussion);
4. No clear distant metastasis at the time of diagnosis of locally recurrent rectal adenocarcinoma or MDT assesses that oligometastatic lesions are resectable or controlable (UICC 8th edition);
5. No previous radiotherapy for initial treatment, or more than 6 months between completion of initial radiotherapy and start of re-radiotherapy, with a previous radiotherapy dose of less than 50.4 Gy, and no grade 3-4 radiotherapy side effects in the small intestine or bladder;
6. ECOG score for performance status is 0-1 (Appendix 1);
7. Peripheral blood cell counts and liver and kidney function within the following acceptable ranges (tested within 15 days before treatment):

   * White blood cell count more than 3.0×10^9/L or neutrophils more than 1.5×10^9/L;

     * Hemoglobin more than 80 g/L; ③ Platelets more than 100×10^9/L; ④ ALT or AST less than 3 times the upper limit of normal; ⑤ Total bilirubin less than 1.5 times the upper limit of normal; ⑥ Creatinine less than 1.5 times the upper limit of normal;
8. No history of other malignant tumors, non-pregnant or lactating patients, participants must use effective contraception during the study and for 6 months after the last treatment;
9. Expected survival more than 12 months.

Exclusion Criteria:

1. Patients with a history of severe allergies to drugs, including platinum-based drugs, 5-FU, LV, and 5-HT3 receptor antagonists;
2. Patients who have participated in or are participating in other clinical trials within 4 weeks of enrollment;
3. Severe electrolyte abnormalities;
4. Presence of gastrointestinal diseases, such as active ulcers in the stomach or duodenum, ulcerative colitis, or unresected tumors that are actively bleeding; or other conditions that may lead to gastrointestinal bleeding or perforation; or unhealed gastrointestinal perforation after surgical treatment;
5. History of arterial thrombosis or deep vein thrombosis within 6 months; evidence of bleeding history or bleeding tendency within 2 months;
6. Pregnant or lactating women or women with a positive pregnancy test before the first medication; or female participants and their partners unwilling to strictly use contraception during the study;
7. Brain metastases with a diameter greater than 3 cm or a total volume greater than 30 cc;
8. Clinical or radiological evidence of spinal cord compression, or tumors within 3 mm of the spinal cord on MRI;
9. History of other active malignant tumors (except for those who have received curative treatment and have been disease-free for over 3 years or in situ cancers that can be cured with adequate treatment);
10. Severe ECG abnormalities, active coronary artery disease, or severe and uncontrolled angina, newly diagnosed angina, or myocardial infarction within 12 months before participating in the study, congestive heart failure of NYHA class II or above;
11. Patients with active infections (fever above 38°C due to infection);
12. Patients with poorly controlled hypercalcemia, high blood pressure, or diabetes;
13. Patients with severe pulmonary diseases (interstitial pneumonia, pulmonary fibrosis, severe emphysema, etc.);
14. Patients with mental disorders affecting clinical treatment or a history of central nervous system diseases;
15. Patients with severe complications (intestinal obstruction, renal failure, liver failure, cerebrovascular disorders, etc.);
16. Any unresolved toxicity from previous treatments that is grade 2 or higher according to CTCAE (excluding anemia, alopecia, skin pigmentation);
17. Any medical condition that is unstable or may affect patient safety and study compliance;
18. Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 2 years

SECONDARY OUTCOMES:
1-year local progression-free survival (LPFS) | 1 year
1-year overall survival (OS) | 1 year
2-year local progression-free survival (LPFS) | 2 years
2-year overall survival (OS) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen H, Louie AV, Higginson DS, Palma DA, Colaco R, Sahgal A. Stereotactic Radiosurgery and Stereotactic Body Radiotherapy in the Management of Oligometastatic Disease. Clin Oncol (R Coll Radiol). 2020 Nov;32(11):713-727. doi: 10.1016/j.clon.2020.06.018. Epub 2020 Jul 24. PMID 32718762
- [Result] Brooks ED, Chang JY. Time to abandon single-site irradiation for inducing abscopal effects. Nat Rev Clin Oncol. 2019 Feb;16(2):123-135. doi: 10.1038/s41571-018-0119-7. PMID 30401936
- [Result] Dorr W, Gabrys D. The Principles and Practice of Re-irradiation in Clinical Oncology: An Overview. Clin Oncol (R Coll Radiol). 2018 Feb;30(2):67-72. doi: 10.1016/j.clon.2017.11.014. Epub 2017 Dec 9. PMID 29233574
- [Result] Dagoglu N, Mahadevan A, Nedea E, Poylin V, Nagle D. Stereotactic body radiotherapy (SBRT) reirradiation for pelvic recurrence from colorectal cancer. J Surg Oncol. 2015 Mar 15;111(4):478-82. doi: 10.1002/jso.23858. Epub 2015 Feb 2. PMID 25644071
- [Result] Susko M, Lee J, Salama J, Thomas S, Uronis H, Hsu D, Migaly J, Willett C, Czito B, Palta M. The Use of Re-irradiation in Locally Recurrent, Non-metastatic Rectal Cancer. Ann Surg Oncol. 2016 Oct;23(11):3609-3615. doi: 10.1245/s10434-016-5250-z. Epub 2016 May 11. PMID 27169769
- [Result] Denost Q, Frison E, Salut C, Sitta R, Rullier A, Harji D, Maillou-Martinaud H, Rullier E, Smith D, Vendrely V; on behalf the GRECCAR Group. A phase III randomized trial evaluating chemotherapy followed by pelvic reirradiation versus chemotherapy alone as preoperative treatment for locally recurrent rectal cancer - GRECCAR 15 trial protocol. Colorectal Dis. 2021 Jul;23(7):1909-1918. doi: 10.1111/codi.15670. Epub 2021 Jun 10. PMID 33843133
- [Result] PelvEx Collaborative. Induction chemotherapy followed by chemoradiotherapy versus chemoradiotherapy alone as neoadjuvant treatment for locally recurrent rectal cancer: study protocol of a multicentre, open-label, parallel-arms, randomized controlled study (PelvEx II). BJS Open. 2021 May 7;5(3):zrab029. doi: 10.1093/bjsopen/zrab029. PMID 34089596
- [Result] Nordkamp S, Voogt ELK, van Zoggel DMGI, Martling A, Holm T, Jansson Palmer G, Suzuki C, Nederend J, Kusters M, Burger JWA, Rutten HJT, Iversen H. Locally recurrent rectal cancer: oncological outcomes with different treatment strategies in two tertiary referral units. Br J Surg. 2022 Jun 14;109(7):623-631. doi: 10.1093/bjs/znac083. PMID 35416250
- [Result] Kusters M, Dresen RC, Martijn H, Nieuwenhuijzen GA, van de Velde CJ, van den Berg HA, Beets-Tan RG, Rutten HJ. Radicality of resection and survival after multimodality treatment is influenced by subsite of locally recurrent rectal cancer. Int J Radiat Oncol Biol Phys. 2009 Dec 1;75(5):1444-9. doi: 10.1016/j.ijrobp.2009.01.015. Epub 2009 Apr 22. PMID 19395199
- [Result] Sun DS, Zhang JD, Li L, Dai Y, Yu JM, Shao ZY. Accelerated hyperfractionation field-involved re-irradiation combined with concurrent capecitabine chemotherapy for locally recurrent and irresectable rectal cancer. Br J Radiol. 2012 Mar;85(1011):259-64. doi: 10.1259/bjr/28173562. Epub 2011 Mar 8. PMID 21385917
- [Result] Rahbari NN, Ulrich AB, Bruckner T, Munter M, Nickles A, Contin P, Loffler T, Reissfelder C, Koch M, Buchler MW, Weitz J. Surgery for locally recurrent rectal cancer in the era of total mesorectal excision: is there still a chance for cure? Ann Surg. 2011 Mar;253(3):522-33. doi: 10.1097/SLA.0b013e3182096d4f. PMID 21209587
- [Result] Yamada K, Ishizawa T, Niwa K, Chuman Y, Akiba S, Aikou T. Patterns of pelvic invasion are prognostic in the treatment of locally recurrent rectal cancer. Br J Surg. 2001 Jul;88(7):988-93. doi: 10.1046/j.0007-1323.2001.01811.x. PMID 11442533
- [Result] Moore HG, Shoup M, Riedel E, Minsky BD, Alektiar KM, Ercolani M, Paty PB, Wong WD, Guillem JG. Colorectal cancer pelvic recurrences: determinants of resectability. Dis Colon Rectum. 2004 Oct;47(10):1599-606. doi: 10.1007/s10350-004-0677-x. PMID 15540287
- [Result] Zhao J, Du CZ, Sun YS, Gu J. Patterns and prognosis of locally recurrent rectal cancer following multidisciplinary treatment. World J Gastroenterol. 2012 Dec 21;18(47):7015-20. doi: 10.3748/wjg.v18.i47.7015. PMID 23323002
- [Result] Westberg K, Palmer G, Hjern F, Johansson H, Holm T, Martling A. Management and prognosis of locally recurrent rectal cancer - A national population-based study. Eur J Surg Oncol. 2018 Jan;44(1):100-107. doi: 10.1016/j.ejso.2017.11.013. Epub 2017 Nov 26. PMID 29224985
- [Result] Lee DJ, Sagar PM, Sadadcharam G, Tan KY. Advances in surgical management for locally recurrent rectal cancer: How far have we come? World J Gastroenterol. 2017 Jun 21;23(23):4170-4180. doi: 10.3748/wjg.v23.i23.4170. PMID 28694657
- [Result] Bouchard P, Efron J. Management of recurrent rectal cancer. Ann Surg Oncol. 2010 May;17(5):1343-56. doi: 10.1245/s10434-009-0861-2. Epub 2009 Dec 30. PMID 20041351
- [Result] Gunderson LL, Jessup JM, Sargent DJ, Greene FL, Stewart A. Revised tumor and node categorization for rectal cancer based on surveillance, epidemiology, and end results and rectal pooled analysis outcomes. J Clin Oncol. 2010 Jan 10;28(2):256-63. doi: 10.1200/JCO.2009.23.9194. Epub 2009 Nov 30. PMID 19949015
- [Result] Hagemans JAW, van Rees JM, Alberda WJ, Rothbarth J, Nuyttens JJME, van Meerten E, Verhoef C, Burger JWA. Locally recurrent rectal cancer; long-term outcome of curative surgical and non-surgical treatment of 447 consecutive patients in a tertiary referral centre. Eur J Surg Oncol. 2020 Mar;46(3):448-454. doi: 10.1016/j.ejso.2019.10.037. Epub 2019 Nov 3. PMID 31761506
- [Result] Sebag-Montefiore D, Stephens RJ, Steele R, Monson J, Grieve R, Khanna S, Quirke P, Couture J, de Metz C, Myint AS, Bessell E, Griffiths G, Thompson LC, Parmar M. Preoperative radiotherapy versus selective postoperative chemoradiotherapy in patients with rectal cancer (MRC CR07 and NCIC-CTG C016): a multicentre, randomised trial. Lancet. 2009 Mar 7;373(9666):811-20. doi: 10.1016/S0140-6736(09)60484-0. PMID 19269519
- [Result] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Result] Swedish Rectal Cancer Trial; Cedermark B, Dahlberg M, Glimelius B, Pahlman L, Rutqvist LE, Wilking N. Improved survival with preoperative radiotherapy in resectable rectal cancer. N Engl J Med. 1997 Apr 3;336(14):980-7. doi: 10.1056/NEJM199704033361402. PMID 9091798
- [Result] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402